CLINICAL TRIAL: NCT06004674
Title: Using Placental Pathology to Prevent Recurrent Adverse Pregnancy Outcomes: A Pilot Project (UPPPP Trial)
Brief Title: Using Placental Pathology to Prevent Recurrent Adverse Pregnancy Outcomes: A Pilot Project
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Sunitha Suresh, Physician, FPA, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EH22-128
Record Dates: First submitted 2023-08-08; First posted 2023-08-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Adverse Pregnancy Outcome
Keywords: miscarriage; preeclampsia; preterm delivery; stillbirth; Low birth weight
MeSH Terms: conditions — Abortion, Spontaneous; Pre-Eclampsia; Premature Birth; Stillbirth | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Placental pathologist will be masked to the outcome when assessing for maternal vascular malperfusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enoxaparin Group (Experimental): Participants in the enoxaparin group will be asked to take a dose of the enoxaparin once a day (40 mg daily) daily from 12 0/7 weeks and/or start of enrollment (whichever is later), and continue until 36 weeks gestational age, after which enoxaparin will be discontinued.
  Interventions: Drug: Lovenox 40mg
- Control Group (No Intervention): Participants in this group will have standard care as usual, with no additional medications.

INTERVENTIONS:
Drug: Lovenox 40mg — Enoxaparin is a blood thinner. It is approved for use in the prevention of deep vein thrombosis (DVT) in abdominal surgery, hip replacement surgery, knee replacement surgery, or medical patients with severely restricted mobility during acute illness; inpatient treatment of acute DVT with or without pulmonary embolism; outpatient treatment of acute DVT without pulmonary embolism; Prevention of ischemic complications of unstable angina and non-Q-wave myocardial infarction; treatment of acute ST-segment elevation myocardial infarction(STEMI) managed medically or with subsequent percutaneous coronary intervention. The use of Lovenox has been shown to be safe, and it has also been used widely off-label in pregnancy.
  Other Names: Enoxaparin
  Arms: Enoxaparin Group

SUMMARY:
The goal of this randomized clinical trial is to evaluate if we can use placental pathology in a prior pregnancy which had an adverse outcome, such as early delivery, stillbirth, a baby born smaller than expected, or severe forms of high blood pressure during pregnancy, to guide treatment in the subsequent pregnancy and reduce risk of recurrent adverse pregnancy events.

The main questions it aims to answer are:

* Whether enoxaparin prevents recurrent adverse pregnancy outcomes among patients with a prior adverse pregnancy outcome that occurred in the setting of maternal vascular malperfusion (MVM).
* If enoxaparin reduces the occurrence or severity of MVM among patients with a prior adverse pregnancy outcome that occurred in the setting of MVM.

DETAILED DESCRIPTION:
In this clinical trial, participants will undergo consent, blood samples will be collected, and participants will be randomized in a 1:1 ratio to the enoxaparin or control groups at their first study visit.

* Participants will return for a study visit within 1 week following randomization.
* If assigned to the enoxaparin, the participant will be asked to take a dose of the enoxaparin once a day (40 mg daily) daily from 12 0/7 weeks and/or the start of enrollment (whichever is later) and continue until 36 weeks gestational age, after which enoxaparin will be discontinued.
* Participants in the control group will have care as usual, with no additional medications.
* During this study, a study team member will collect a blood sample from all participants at 20-24 weeks, 32-34 weeks, and at delivery.
* Participants in the enoxaparin group will have their blood work checked a week after starting medication to ensure that they have no unanticipated side effects.

Researchers will compare the enoxaparin group to the control group to see if enoxaparin prevents or reduces the occurrence or severity of maternal vascular malperfusion (MVM) among patients with a prior adverse pregnancy outcome.

ELIGIBILITY:
Eligibility Criteria:

Inclusion (must meet all three criteria):

1. Subjects with a prior adverse outcome in a prior pregnancy. Adverse outcome is defined as prior singleton preterm birth ( < 37 weeks), SGA infant (defined as birthweight < 10th percentile), preeclampsia with severe features, or stillbirth (fetal demise after 20 weeks gestation), as certified by an obstetrician
2. Patients with maternal vascular malperfusion on pathology from pregnancy with prior adverse pregnancy outcome, as certified by a perinatal placental pathologist
3. Current singleton pregnancy at <16 6/7 weeks gestational age.

Exclusion Criteria:

1. Anticoagulation planned for current pregnancy (including warfarin, enoxaparin, heparin)
2. Known major fetal anomaly
3. Contraindication to enoxaparin: Specifically active major bleeding, known thrombocytopenia (platelets <100), hypersensitivity to enoxaparin sodium, hypersensitivity to heparin or pork products, hypersensitivity to benzyl alcohol
4. Chronic kidney disease with eGFR< 60
5. Known chronic liver disease with baseline AST/ALT > 3 x upper limit of normal
6. Subjects with mechanical prosthetic heart valves

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study will specifically recruit patients who are pregnant, and we anticipate that they will primarily be of female sex.
Enrollment: 20 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Composite Adverse Pregnancy outcome | Enrollment through 6 weeks postpartum
  Preeclampsia with severe features, small for gestational age infant, preterm delivery <37 weeks, neonatal death, and maternal death

SECONDARY OUTCOMES:
Maternal vascular malperfusion (MVM) | Placenta collected at time of delivery
  Presence/ absence of MVM on placental pathology
Preeclampsia with severe features | Enrollment through 6 weeks postpartum
  Defined by clinician
Small for gestational age infant | At time of delivery
  By Fenton criteria
Preterm delivery < 37 weeks | Assessed at time of delivery
Neonatal Death | Assessed from time of delivery to 6 weeks postpartum
Maternal Death | Assessed from enrollment to 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha Suresh, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No